CLINICAL TRIAL: NCT02936037
Title: Effect of MD1003 in Progressive Multiple Sclerosis: a Randomized Double Blind Placebo Controlled Study
Brief Title: Effect of MD1003 in Progressive Multiple Sclerosis (SPI2)
Acronym: SPI2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision for business purposes
Sponsor: MedDay Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MD1003CT2016-01MS-SPI2
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Multiple Sclerosis
Keywords: progressive multiple sclerosis; MS; EDSS; TW25; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Biotin

STUDY DESIGN:
Intervention Model Description: PART 1:
  Total duration of Part 1 is 27 months. The randomized double-blind placebo-controlled period ranges from 15 to 27 months depending upon the randomization date of an individual patient.
  Once the last month 15 evaluation of the study has been completed, patients will switch to the active drug at the next planned visit. Participants and study personnel will remain blinded as to the original treatment assignment.
  Maximum duration of double-blind period per patient will be no longer than 27 months.
  PART 2:
  At the last evaluation of Part 1 (Visit 11/Month 27) all participants will be offered active treatment in an open label extension for 39 additional months (From V11/M27 to V18/M66).
  The purpose of the active drug extension is to further define the safety of MD1003.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GROUP 1 (Placebo Comparator): Placebo capsule, 1 capsule tid (morning,noon and evening) for 15 months and up to 27 months.
  Interventions: Drug: PLACEBO
- GROUP 2 (Experimental): MD1003 capsule, 1 capsule tid (morning,noon and evening) for 15 months and up to 27 months.
  Interventions: Drug: MD1003 100mg capsule

INTERVENTIONS:
Drug: MD1003 100mg capsule
  Other Names: high dose biotin
  Arms: GROUP 2
Drug: PLACEBO — an inactive substance
  Arms: GROUP 1

SUMMARY:
The purpose of this study is to demonstrate the superiority of MD1003 over placebo in the disability of patients suffering from progressive multiple sclerosis and especially those with gait impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-65 years old
* Signed and dated written informed consent form in accordance with local regulations: having freely given their written informed consent to participate in the study
* Diagnosis of primary or secondary progressive MS fulfilling revised McDonald criteria (2010) and Lublin criteria (2014)
* Documented evidence of clinical disability progression within the 2 years prior to inclusion, i.e. a) progression of EDSS during the past two years of at least 1 point sustained for at least 6 months if inclusion EDSS is from 3.5 to 5.5 or at least 0.5 point increase sustained for at least 6 months if inclusion EDSS is from 6 to 6.5 or b) increase of TW25 by at least 20% in the last two years sustained for at least 6 months or c) other well-documented objective worsening validated by the Adjudication Committee
* EDSS at inclusion from 3.5 to 6.5
* TW25 < 40 seconds at inclusion visit
* Kurtzke pyramidal functional subscore ≥2 defined as "minimal disability: patient complains of motor-fatigability or reduced performance in strenuous motor tasks (motor performance grade 1) and/or BMRC grade 4 in one or two muscle groups"

Exclusion Criteria:

* Clinical evidence of a relapse in 24 months prior to inclusion
* Treatment with any product containing biotin as single ingredient within six months prior to inclusion (multivitamin supplementation authorized if biotin < 1mg per day)
* Concomitant treatment with fampridine at inclusion or in the 30 days prior to inclusion
* New immunosuppressive/immunomodulatory drug initiated less than 90 days prior to inclusion
* Treatment with botulinum toxin (except for cosmetic purpose) initiated within 6 months prior to inclusion
* In-patient rehabilitation program within the 3 months prior to inclusion
* Pregnancy, breastfeeding or women with childbearing potential without acceptable form of contraception
* Men unwilling to use an acceptable form of contraception
* Any general chronic handicapping/incapacitating disease other than MS
* Any serious disease necessitating biological follow-up with biological tests using biotinylated antibodies or substrates
* Past history of rhabdomyolysis/metabolic myopathy
* Known fatty acids beta oxidation defect
* Known hypersensitivity or intolerance to biotin, analogues or excipients, patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Patients with hypersensitivity or any contra-indication to Gadolinium
* Patients with uncontrolled hepatic disorder, renal or cardiovascular disease, or cancer
* Laboratory tests out of normal ranges considered by the investigator as clinically significant with regards to the study continuation
* Patients with history or presence of alcohol abuse or drug addiction
* Untreated or uncontrolled psychiatric disorders, especially suicidal risk assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
* Participation in another research study involving an investigational product (IP) in the 90 days prior to inclusion, or planned use during the study duration
* Patients likely to be non-compliant to the study procedures or for whom a long-term follow-up seems to be difficult to achieve
* Relapse that occurs between inclusion and randomization visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Cree, MD, PHD, Principal Investigator — University of California, San Francisco; Frederic Sedel, MD, PHD, Study Director — Medday Pharmaceuticals
Locations (92):
- United States (40):
  - Barrow Neurology Clinics (BNC), Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Jordan Research And Education Institute Of Alta Bates Summit, Berkeley, California
  - Neuro-Pain Medical Center, Fresno, California
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - MS Center of California, Newport Beach, California
  - UC Davis Health System, Sacramento, California
  - UCSF Multiple Sclerosis Center, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale New Haven Hospital, North Haven, Connecticut
  - Nova Clinical Research, LLC, Bradenton, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of South Florida - Neurology, Tampa, Florida
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago Medical Center-Duchossois Center for Advanced Medicine (DCAM), Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Rowe Neurology Institute, Lenexa, Kansas
  - Ochsner Health System, New Orleans, Louisiana
  - The Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Harvard Medical School - Brigham and Women's Hospital - Center for Neurologic Diseases, Boston, Massachusetts
  - Wayne State University - Comp Clinic and MS Center, Detroit, Michigan
  - Minneapolis Clinic of Neurology, LTD, Golden Valley, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Holy Name Hospital, Teaneck, New Jersey
  - The University of New Mexico - Multiple Sclerosis Specialty Clinic, Albuquerque, New Mexico
  - UBMD Neurology, Buffalo, New York
  - Mount Sinai School of Medicine - Corinne Goldsmith Dickinson Center for MS, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - State University of New York (SUNY), Stony Brook, New York
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - Cleveland Clinic Mellen Center for MS, Cleveland, Ohio
  - Providence Multiple Sclerosis Center, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Vanderbilt Comprehensive Multiple Sclerosis Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Australia (3):
  - Brain and Mind Centre/University of Sydney, Sydney, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Belgium (3):
  - UZ Antwerpen, Edegem, Antwerpen
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt, Limburg
  - UZ Gent, Halle, Oost-Vlaanderen
- Canada (8):
  - Burnaby Hospital, Burnaby, British Columbia
  - Vancouver Hospital and Health Sciences Centre, Vancouver, British Columbia
  - Hôpital universitaire Dr George L-Dumont university Hospital, Moncton, New Brunswick
  - Nova Scotia Rehabilitation Center, Halifax, Nova Scotia
  - Ottawa Hospital General Campus, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Hopital de Notre Dame, Montreal, Quebec
  - Montreal Neurologic Institute, Montreal, Quebec
- Czechia (5):
  - doc. MUDr. Radomir Talab, CSc., neurologie, Hradec Králové
  - Nemocnice Jihlava, Jihlava
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
  - Nemocnice Teplice, Teplice
- Germany (10):
  - Universitätsklinikum Leipzig A.ö.R. - Klinik und Poliklinik, Leipzig, Saxony
  - Fachkrankenhaus Hubertusburg, Wermsdorf, Saxony
  - Caritas Krankenhaus, Bad Mergentheim
  - Charité - Universitätsmedizin Berlin / NeuroCure Clinical Research Center, Berlin
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf
  - Neuro Centrum Science GmbH, Erbach im Odenwald
  - MultipEL Studies Institut für klinische Studien GbR, Hamburg
  - Ludwig-Maximilians Universität München, München
  - Neuropoint GmbH, Ulm
  - Poliklinik für Neurologie Universitätsklinikum Ulm, Ulm
- Valeomed Kft, Esztergom, Hungary
- Italy (2):
  - Ospedale San Raffaele, IRCCS, Milan
  - AO S.Andrea, Università degli Studi di Roma La Sapienza, Roma
- Poland (4):
  - Nasz Lekarz Ośrodek Badań Klinicznych, Bydgoszcz
  - COPERNICUS PL sp z o.o.,Szpital im. M.Kopernika Oddział Neurologiczny, Gdansk
  - Twoja Przychodnia Centrum Medyczne Nowa Sol, Nowa Sól
  - Centrum Medyczne Pratia Warszawa, Warsaw
- Spain (7):
  - Hospital Santa Caterina, Salt, Girona
  - Hostipal Universitario Quirónsalud Madrid, Pozuelo de Alarcón, Madrid
  - Servicio de Neurología Hospital Vithas Nisa Aljarafe, Castilleja de la Cuesta, Sevilla
  - Hospital del Mar Servicio de Neurología, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- Sweden (2):
  - Sahlgrenska Universitetssjukhus - MS Center forskningsenheten, Gothenburg
  - Karolinska University Hospital - Neurologmottagningen, Stockholm
- Ondokuz Mayis University Medical Faculty, Samsun, Turkey (Türkiye)
- United Kingdom (6):
  - The University of Edinburgh, Edinburgh
  - Institute of Neurological Sciences, Glasgow
  - Barts And The London School Of Medicine And Dentistry Institute, London
  - University College London Institute of Neurology / National Hospital for Neurology & Neurosurgery, London
  - Tyne Hospitals NHS Foundation, Newcastle upon Tyne
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cree BAC, Cutter G, Wolinsky JS, Freedman MS, Comi G, Giovannoni G, Hartung HP, Arnold D, Kuhle J, Block V, Munschauer FE, Sedel F, Lublin FD; SPI2 investigative teams. Safety and efficacy of MD1003 (high-dose biotin) in patients with progressive multiple sclerosis (SPI2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Neurol. 2020 Dec;19(12):988-997. doi: 10.1016/S1474-4422(20)30347-1. Epub 2020 Oct 23. PMID 33222767

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo capsule, 1 capsule tid (morning,noon and evening) for 15 months and up to 27 months.
  PLACEBO: an inactive substance
- MD1003: MD1003 capsule, 1 capsule tid (morning,noon and evening) for 15 months and up to 27 months.
  MD1003 100mg capsule
Period: Double-Blind Treatment Period
Arm/Group | Placebo | MD1003
Started | 316 | 326
Completed | 267 | 261
Not Completed | 49 | 65
Not completed — Protocol Violation | 1 | 4
Not completed — Suicidal risk, etc. | 2 | 8
Not completed — Lack of Efficacy | 4 | 12
Not completed — Death | 0 | 1
Not completed — Adverse Event | 11 | 11
Not completed — Withdrawal by Subject | 31 | 28
Not completed — Lost to Follow-up | 0 | 1
Period: Open Label Extension
Arm/Group | Placebo | MD1003
Started | 0 | 528
Completed | 0 | 518
Not Completed | 0 | 10
Not completed — Adverse Event | 0 | 3
Not completed — Other | 0 | 3
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MD1003 | Total
Number analyzed (Participants) | 316 | 326 | 642
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (7.60) | 52.6 (7.79) | 52.7 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 175 | 345
  Male | 146 | 151 | 297
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 21
  Not Hispanic or Latino | 293 | 302 | 595
  Unknown or Not Reported | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 8 | 21
  White | 291 | 306 | 597
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  Hungary | 0 | 1 | 1
  United States | 109 | 109 | 218
  Czechia | 26 | 31 | 57
  United Kingdom | 31 | 30 | 61
  Spain | 30 | 31 | 61
  Canada | 35 | 37 | 72
  Sweden | 9 | 9 | 18
  Turkey | 2 | 2 | 4
  Belgium | 4 | 7 | 11
  Poland | 11 | 12 | 23
  Italy | 5 | 7 | 12
  Australia | 6 | 8 | 14
  Germany | 48 | 42 | 90

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Improved on Either Expanded Disability Status Scale (EDSS) or Time to Walk 25 Feet (TW25)
Description: Proportion of patients improved on either Expanded Disability Status Scale (EDSS) or time to walk 25 feet (TW25) :
  - with decreased EDSS at M12 confirmed at M15 (where decreased EDSS is defined as a decrease of at least 1 point if initial EDSS from 3.5 to 5.5 and of at least 0.5 point if initial EDSS from 6 to 6.5)
  or
  - with improved TW25 of at least 20% at Month 12 and Month15
  compared to the lowest of the two EDSS and TW25* scores among inclusion and randomization visits.
  *The lowest TW25 value recorded among the four values obtained during the inclusion and randomization visits will be considered as the baseline TW25 value.
Time Frame: 15 months
Measure: Number; unit: percent
Arm/Group | Placebo | MD1003
Number analyzed (Participants) | 316 | 326
percent | 9.2 | 12.0

2. Secondary Outcome: Time to 12-Weeks Confirmed EDSS Progression
Description: 12-weeks EDSS progression is defined by an increase of at least 1 point for baseline EDSS 3.5 to 5.5 and of at least 0.5 point for baseline EDSS 6 to 6.5 with respective confirmation 12 weeks later.
  Date of 12-weeks confirmed EDSS progression will be the first date of an EDSS progression (as defined above) that is confirmed 12 weeks later.
Time Frame: 3 to 27 months
Reporting Status: Not Posted

3. Secondary Outcome: CGI-I Score (Clinical Global Impression of Change - Improvement), Evaluated Both by the Patient (SGI) and by the Evaluating Physician (CGI)
Time Frame: 15 months
Reporting Status: Not Posted

4. Secondary Outcome: Mean Change in TW25 Between M0 and M15
Time Frame: 15 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Brain MRI Changes Between M0 and M15
Time Frame: 15 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Remote Monitoring of Ambulation
Time Frame: 27 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: (MSQOL54) & (CAREQOL-MS) Subscores and Composite Scores
Time Frame: 15 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Subscores of the Kurtzke Functional Score
Time Frame: 15 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Symbol Digit Modalities Test (SDMT)
Time Frame: 15 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 27 months for the double-blind period, and was to be collected for 39 months in open-label extension before premature termination of the study.
Groups:
- GROUP 2: MD1003 capsule, 1 capsule tid (morning,noon and evening) for 15 months and up to 27 months.
  MD1003 100mg capsule
Arm/Group | GROUP 1 | GROUP 2
All-Cause Mortality (participants affected / at risk) | 0/311 | 1/331
Serious Adverse Events (participants affected / at risk) | 82/311 | 87/331
Other Adverse Events (participants affected / at risk) | 264/311 | 277/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GROUP 1 (N=311) | GROUP 2 (N=331)
Multiple sclerosis relapse (Nervous system disorders) | 31 (37) | 29 (36)
Multiple sclerosis (Nervous system disorders) | 6 (7) | 4 (4)
Trigeminal neuralgia (Nervous system disorders) | 4 (4) | 1 (1)
Muscle spasticity (Nervous system disorders) | 1 (1) | 3 (3)
Uhthoff's phenomenon (Nervous system disorders) | 1 (2) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Sensory Loss (Nervous system disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Cataplexy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Facial spasm (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Narcolepsy (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Pyramidal tract syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Transverse sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (6) | 2 (3)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Urosepsis (Infections and infestations) | 3 (3) | 2 (2)
Bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Haemorrhagic pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Human anaplasmosis (Infections and infestations) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diaphragmatic hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Breathing-related sleeping disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Silent myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cystadenocarcinoma ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Elective procedure (Surgical and medical procedures) | 1 (1) | 1 (1)
Neurological rehabilitation (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastric banding reversal (Surgical and medical procedures) | 0 (0) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Factor V Leiden mutation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Device failure (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GROUP 1 (N=311) | GROUP 2 (N=331)
Urinary tract infection (Infections and infestations) | 50 (94) | 48 (74)
Nasopharyngitis (Infections and infestations) | 58 (76) | 39 (53)
Upper respiratory tract infection (Infections and infestations) | 27 (34) | 25 (33)
Multiple sclerosis relapse (Nervous system disorders) | 31 (37) | 29 (36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (31) | 25 (29)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 24 (33) | 20 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (21) | 19 (25)
Fall (Injury, poisoning and procedural complications) | 37 (60) | 44 (84)
Contusion (Injury, poisoning and procedural complications) | 23 (26) | 13 (20)
Constipation (Gastrointestinal disorders) | 16 (16) | 18 (19)
Fatigue (General disorders) | 26 (28) | 24 (26)
Gait disturbance (General disorders) | 17 (21) | 22 (28)
Laboratory test interference (Investigations) | 1 (1) | 25 (28)
Depression (Psychiatric disorders) | 12 (12) | 17 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT02936037/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT02936037/SAP_001.pdf